CLINICAL TRIAL: NCT05220384
Title: Motivational, Movement and Self-Management Training for Hungarian Adolescents Living With Chronic Pain
Brief Title: Motivational, Movement and Self-Management Training for Adolescents in Pain
Acronym: M3 Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IV/7741-3/2021/EKU
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; self-management; adolescent; motivation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized In-person therapy (Other)
  Interventions: Behavioral: In-person Motivational Interview combined with Self-Management techniques
- Generalized, Video-based therapy (Other)
  Interventions: Behavioral: Video-based Motivational Interview combined with Self-Management techniques

INTERVENTIONS:
Behavioral: In-person Motivational Interview combined with Self-Management techniques — This is an approximately 30 mins in-person, semi-structured, semi-personalized physical activity focused Motivational Interviewing treatment with self-management techniques. (This therapy is an add on to the "usual therapy" that is given to the adolescents who present at the hospital.) During the interactive treatment a self-management workbook will be filled out by the adolescent for the purpose of further data collection. This in-person therapy at the hospital is followed by two booster sessions via phone at the 1st week post meeting date and 1 month post meeting date.
  Arms: Personalized In-person therapy
Behavioral: Video-based Motivational Interview combined with Self-Management techniques — This is a series of three videos comprising a structured activity focused Motivational Interviewing treatment with self-management techniques. The videos' thematic follow the semi-structured interview elements to ensure that it is a true sham of the in-person one. (This therapy is an add on to the "usual therapy" that is given to the adolescents who present at the hospital.) This first video is going to be watched by adolescents at the hospital. During the interactive video-treatment a self-management workbook will be filled out by the adolescent for the purpose of further data collection. The second video is going to be sent to the participants via e-mail on the 1st week post meeting date and the third video is on the 1-month post meeting date.
  Arms: Generalized, Video-based therapy

SUMMARY:
With this randomized controlled trial, we have three aims. First of all, to investigate underlying mechanisms that might contribute to the success of a physical activity focused self-management program in paediatric chronic pain.

Second of all, to determine the minimum intervention needed for improving physical activity amongst adolescents who live with chronic pain. For this we are comparing an in-person and a video-based motivational interviewing training combined with self-management techniques.

Third of all, to investigate the mediating effect of autonomy in adolescents with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-18 years
* Experiencing pain at least 3 months
* Good reading, writing and listening skills in Hungarian language
* Self-sufficient
* Access to internet and phone
* No active cancer.

Exclusion Criteria:

* Age is not between 12-18 years
* Experiencing pain less then 3 months
* Not able to read, write and listen in Hungarian
* Not self-sufficient
* No access to internet and phone
* Active cancer.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Child Self-Efficacy Scale | 3 months
  The Pain Self-efficacy Scale is a 7item measure assessing child self-efficacy for functioning normally when in pain (PSES-C, PSES-P; Bursch et al., 2006). An example item is "How sure are you that you can take care of yourself when you have pain?" Items are scored on a 5-point Likert scale with lower scores indicating higher self-efficacy. Initial validation provided support for the measure's validity and reliability, and internal consistency in this sample was strong (a ¼ .90).

SECONDARY OUTCOMES:
Visual Analog Scale | 3 months
  Pain Intensity cores were anchored at 0="no pain" to 100="unbearable pain", with higher scores reflecting greater pain intensity.
Revised Children's Anxiety and Depression Scale | 3 months
  Depression, Anxiety The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item, youth self-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Additionally, The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) similarly assesses parent report of youth's symptoms of anxiety and depression across the same six subscales.
State-Trait Anxiety Inventory for Children | 3 months
  Anxiety The STAI-CH is the definitive instrument for measuring anxiety in children. Based on the same theory as the STAI, the State-Trait Anxiety Inventory for Children (STAI-CH) distinguishes between a general proneness to anxious behavior rooted in the personality and anxiety as a fleeting emotional state. The instrument is designed to be used with upper elementary or junior high school aged children and consists of two twenty-item scales. The measure is easy to read and can be administered verbally to younger children.
Paediatric Pain Disability Index | 3 months
  Disability Each of the 7 items is rated on a scale from 0 to 10 where 0 means no disability and 10 means total disability.
  PDI results range from 0 to 70 where the higher the score, the greater the degree of disability and impact on life activities due to pain.
  The PDI is used for initial evaluations and for monitoring pain relief effectiveness and response to other interventions.
Pain Stages of Change Questionnaire for Adolescents and for Parents | 3 months
  Readiness to change The 30-item PSOCQ-A and -P measures include parallel items rated on a 5-point scale: 1="Strongly Disagree", 2="Disagree", 3="Undecided or Unsure", 4="Agree", 5="Strongly Agree". Greater readiness to change was conceptualized as lower Precontemplation and/or higher Action/Maintenance scores, while less readiness to change was represented by higher Precontemplation and/or lower Action/Maintenance scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Health Services Management Training Centre, Budapest, Pest State, Hungary

IPD SHARING:
Plan to Share IPD: Undecided